CLINICAL TRIAL: NCT02515747
Title: Role of Lipoprotein(a) Concentration and Apolipoprotein(a) Phenotype in Prediction of Coronary Events in General Population
Brief Title: Prospective Russian Evaluation of Lp(a) Role in cardiovascUlar DiseasE
Acronym: PRELUDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Cardiology Research and Production Center (Other)
Responsible Party: Principal Investigator, Marat Vladislavovich Ezhov (MV Ezhov, MD, PhD, DMSc), Associate Professor, Dr., Russian Cardiology Research and Production Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01200406198
Record Dates: First submitted 2015-05-08; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Disease; Cardiovascular Diseases
Keywords: Lipoprotein(a); coronary artery bypass grafting (CABG); apo(a); prognosis; myocardial infarction; cardiovascular death; percutaneous coronary intervention (PCI)
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Myocardial Infarction | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- conservative treatment (No Intervention): Men and women with stable CHD verified by angiography from one center and allocated to three treatment arms in real-world practice: 1. conservative treatment with statins, antiaggregants, antianginal drugs in standard dosage
- percutaneous coronary intervention (Active Comparator): 2. elective balloon angioplasty alone or stent implanation on the basement of drugs treatment
  Interventions: Procedure: percutaneous coronary intervention
- coronary artery bypass grafting (Active Comparator): elective surgery myocardial revascularisation on the basement of drugs treatment
  Interventions: Procedure: coronary artery bypass grafting

INTERVENTIONS:
Procedure: percutaneous coronary intervention — elective percutaneous coronary balloon angioplasty and/or stenting
  Arms: percutaneous coronary intervention
Procedure: coronary artery bypass grafting — elective surgical myocardial revascularisation
  Arms: coronary artery bypass grafting

SUMMARY:
The purpose of this study is to explore the role of lipoprotein(a) and apolipoprotein(a) phenotype in fatal and non-fatal cardiovascular disease (CVD) events risk in coronary disease patients divided on the basis of management strategy - medical, endovascular or open cardiac surgery.

DETAILED DESCRIPTION:
Between January 1993 and September 2006, we enrolled 1400 consecutive patients from the Atherosclerosis Department with known Lp(a) levels and coronary heart disease (CHD) verified by angiography. In accordance with clinical condition and angiography data were assigned them into three parallel treatment arms and followed up to 15 years. This study was conducted according to the principles of the Declaration of Helsinki and the Institutional Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* stable coronary heart disease verified by angiography

Exclusion Criteria:

* acute coronary syndromes,
* acute infections,
* inflammatory disease within 3 months prior to inclusion,
* familial hypercholesterolemia,
* triglycerides>4.5 mmol/L,
* missing Lp(a) measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 1993-01; Primary Completion 2006-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
non-fatal myocardial infarction and cardiovascular death | up to 15 years
  we took a composite primary outcome measure because anticipated a low number of hard-end-points in each treatment arm

SECONDARY OUTCOMES:
non-fatal myocardial infarction and cardiovascular death and myocardial revascularisation and hospitalization for recurrent or unstable angina | up to 15 years
  we chose a composite secondary outcome mesure as a standard for such type studies and to obtain a statistical difference between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Marat V. Ezhov, PhD, DMSc, Principal Investigator — Russian Cardiology Research and Production Center; Sergei N. Pokrovsky, PhD, DSc, Study Chair — Russian Cardiology Research and Production Center; Valery V. Kukharchuk, PhD, DMSc, Study Chair — Russian Cardiology Research and Production Center

REFERENCES:
- [Background] Ezhov MV, Afanas'eva OI, Kambegova AA, Afanas'eva MI, Trukhacheva EP, Naumov VG, Pokrovskii SN. [The role of atherosclerosis risk factors in development of ischemic heart disease in young men]. Ter Arkh. 2009;81(5):50-4. Russian. PMID 19537587
- [Background] Ezhov MV, Liakishev AA, Pokrovskii SN. [Lipoprotein (a) - an independent risk factor in atherosclerosis]. Ter Arkh. 2001;73(9):76-82. No abstract available. Russian. PMID 11642088
- [Result] Pokrovsky SN, Ezhov MV, Il'ina LN, Afanasieva OI, Sinitsyn VY, Shiriaev AA, Akchurin RS. Association of lipoprotein(a) excess with early vein graft occlusions in middle-aged men undergoing coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2003 Oct;126(4):1071-5. doi: 10.1016/s0022-5223(03)00365-9. PMID 14566249
- [Result] Ezhov MV, Safarova MC, Afanas'eva OI, Il'ina LN, Liakishev AA, Pokrovskii SN. [High level of lipoprotein (a) as a predictor of poor long-term prognosis after coronary artery bypass surgery]. Kardiologiia. 2011;51(1):18-22. Russian. PMID 21626797
- [Result] Ezhov MV, Safarova MS, Afanasieva OI, Kukharchuk VV, Pokrovsky SN. Lipoprotein(a) level and apolipoprotein(a) phenotype as predictors of long-term cardiovascular outcomes after coronary artery bypass grafting. Atherosclerosis. 2014 Aug;235(2):477-82. doi: 10.1016/j.atherosclerosis.2014.05.944. Epub 2014 Jun 4. PMID 24952151
- [Result] Britareva VV, Afanas'eva OI, Dobrovol'skii AB, Ezhov MV, Titaeva EV, Karpov IuA, Pokrovskii SN. [Lipoprotein(a) and Apo-A isoforms in patients with intermittent claudication]. Ter Arkh. 2002;74(12):49-52. Russian. PMID 12577841
- [Result] Ezhov MV, Afanas'eva OI, Benevolenskaia GF, Savchenko AP, Balakhonova TV, Liakishev AA, Pokrovskii SN. [Association of lipoprotein(a) and apolipoprotein(a) phenotypes with coronary and carotid atherosclerosis in CHD men]. Ter Arkh. 2000;72(1):28-32. Russian. PMID 10687202
- [Result] Ezhov MV, Afanas'ev OI, Benevolenskaia GF, Savchenko AP, Liakishev AA, Pokrovskii SN. [Lipoprotein(a) as a biochemical marker of coronary atherosclerosis]. Ter Arkh. 1997;69(9):31-4. Russian. PMID 9411822
- [Result] Safarova MS, Trukhacheva EP, Ezhov MV, Afanas'eva OI, Afanas'eva MI, Tripoten' MI, Liakishev AA, Pokrovskii SN. [Pleiotropic effects of nicotinic acid therapy in men with coronary heart disease and elevated lipoprotein(a) levels]. Kardiologiia. 2011;51(5):9-16. Russian. PMID 21649590